CLINICAL TRIAL: NCT04957004
Title: Evaluation of Left Ventricular Function and Therapeutic Effect of CPAP in Patients With OSAS by 3D Speckle-tracking Echocardiography
Brief Title: Evaluation of Left Ventricular Function and Therapeutic Effect of CPAP in Patients With OSAS by 3D STE
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2017397
Record Dates: First submitted 2021-06-29; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: OSA; Left Ventricular Dysfunction
Keywords: OSA; CPAP; left ventricular dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OSA patients: Patients with OSA who have not been treated with CPAP
  Interventions: Device: CPAP
- control group: health control except OSA by using sleep monitorin

INTERVENTIONS:
Device: CPAP — CPAP ventilator was worn at nigh
  Groups: OSA patients

SUMMARY:
The changes of left ventricular function in patients with sleep apnea were studied by three-dimensional speckle-tracking echocardiography to evaluate the changes of left ventricular function after CPAP treatment

DETAILED DESCRIPTION:
Research purposes: (1) Use 3D speckle tracking echocardiography to measure the diastolic and systolic strains of the left atrium and left ventricle of OSAS patients, in order to evaluate the impact and degree of OSA on left ventricular function.

(2) By comparing the changes in the three-dimensional ultrasound strain index of the left ventricle of patients before and after CPAP treatment, and in patients receiving and not receiving CPAP treatment, to evaluate whether CPAP treatment contributes to the improvement of cardiac function in patients with OSAS, and to infer the best suitable intervention population and using time, providing reference basis for clinical treatment.

(3) Discovery of serological indicators that predict the severity of the disease and predict the impairment of heart function Study design: This study is a prospective, observational controlled study. It is planned to include 30 cases of newly diagnosed OSAS patients in the Peking University Third Hospital and a control group selected according to age and gender matching. The three-dimensional strain of the left atrium and left ventricle of the crowd is measured by the 3D speckle tracking technology, and the serological indicators are detected. The OSAS group and the control group were followed up during the course of receiving or not receiving CPAP.

ELIGIBILITY:
Inclusion Criteria:

1. OSA met the diagnostic criteria of obstructive sleep apnea in the United States Classification of Sleep Diseases in 2014
2. Between the ages of 18 and 80, regardless of gender
3. Sign informed consent

Exclusion Criteria:

1. previously diagnosed patients with heart failure,
2. coronary artery disease,
3. valvular disease,
4. cardiomyopathy,
5. arrhythmia,
6. chronic obstructive/ restrictive pulmonary disease,
7. thyroid dysfunction (including hypothyroidism or hyperthyroidism),
8. already treated with CPAP,
9. poor image quality of echocardiography.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with OSA who underwent sleep monitoring at the Sleep Medicine Center of Peking University Third Hospital were selected for the study.OSA met the diagnostic criteria of obstructive sleep apnea in the United States Classification of Sleep Diseases in 2014.Exclusion criteria from this study included previously diagnosed patients with heart failure,coronary artery disease,valvular disease,cardiomyopathy,arrhythmia,chronic obstructive/ restrictive pulmonary disease, thyroid dysfunction (including hypothyroidism or hyperthyroidism), already treated with CPAP, and poor image quality of echocardiography. Healthy subjects who underwent sleep monitoring to exclude OSA were selected as the control group during the same period.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-07-22 (Actual); Primary Completion 2019-12-22 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
The changes of echocardiographic and serological indexes were observed by 3D speckled tracking during the 1-year follow-up | The follow-up period was 1 year
  The changes of echocardiographic indexs such as left ventricular three-dimensional strain and serological indexes including adiponectin.

CONTACTS AND LOCATIONS:
Overall Officials: Yongzhen Zhang, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No